CLINICAL TRIAL: NCT03423420
Title: High Central Venous Pressure After Cardiac Surgery is Associated With Increased Morbidity and Mortality
Brief Title: Pontos-Central Venous Pressure and Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Felix Balzer, Prof. Dr. med. Dr. rer. nat., MSc, Charite University, Berlin, Germany
Other Study IDs: PONTOS-CVP
Record Dates: First submitted 2018-01-25; First posted 2018-02-06 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Central Venous Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Recent studies indicated the central venous pressure (CVP) as a prognostic marker. Therefore, we retrospectively analyzed the CVP on admission to the intensive care unit (ICU) in cardiac surgery patients regarding its prognostic value for morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* In-patients of the Charité Universitätsmedizin Berlin
* at least 18 years old
* female or male sex
* cardiosurgical intervention (OPS 5.35 and 5.36) between 01/06 and 12/13.
* post-operative monitoring of anesthesiological intensive care unit

Exclusion Criteria:

* previous cardiosurgical interventions during the same hospital stay.
* incomplete documentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult male and female patients who have undergone cardiac surgery in the period 01/06-12/13 at Campus Mitte in the Charité, approx. 7000 patients.
Sampling Method: Probability Sample
Enrollment: 5945 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
mortality | an average of 30 days
  In-Hospital mortality

SECONDARY OUTCOMES:
Central venous pressure | intensive care unit stay, an average of 5 days
  central venous pressure on intensive care unit
Hospital stay | an average of 13 days
  Length of hospital stay
ICU stay | an average of 5 days
  Intensive care unit length of stay
ICU readmission | an average of 30 days
  Amount of hospital readmissions
Renal insufficiency - 1 | intensive care unit stay, an average of 5 days
  Incidence of renal insufficiency
Renal insufficiency - 2 | intensive care unit stay, an average of 5 days
  dialysis duration
Renal insufficiency - 3 | intensive care unit stay, an average of 5 days
  Urine production
Stroke | hospital length of stay, an average of 13 days
  incidence of strokes
mortality rate-1 | 90 days
  mortality rate after 90 days
mortality rate-2 | 180 days
  mortality rate after 180 days
mortality rate-3 | 3 years
  mortality rate after 3 years
mortality rate-4 | 1 year
  mortality rate after 1 year
mortality rate-5 | 5 years
  mortality rate after 5 years

OTHER OUTCOMES:
priority of surgery | an average of 1 day
  priority of surgery selected from a three point categorial scale with the categories elective, urgent and emergency
type of surgery | an average of 1 day
  type of surgery selected from the three point categorial scale with categories bypass graft, valve replacement or combination of both
duration | an average of 4 hours
  duration of surgery
APACHE II | an average of 30 days
  APACHE II Score of patients on admission on the ICU
ACEF Score | an average of 1 day
  preoperative ACEF Score of patients undergoing surgery

CONTACTS AND LOCATIONS:
Overall Officials: Felix Balzer, MD, MSc, PhD, Principal Investigator — Charite Universitätsmedizin Berlin
Locations (1):
- Charité - Universitaetsmedizin Berlin, Berlin, Germany